CLINICAL TRIAL: NCT07248553
Title: The Effect of Levonorgestrel-Containing Intrauterine Device (LNG-IUD) Insertion Timing on Ovarian Cyst Development According to the Early and Late Follicular and Luteal Phases
Brief Title: Timing of LNG-IUD Insertion and Ovarian Cyst Formation
Acronym: LNG-IUD TIMING
Status: Recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Betül Bacak, Specialist in Obstetrics and Gynecology, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GOPEAH-LNGIUD
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cysts; Menstrual Cycle; Intrauterine Device (IUD)
Keywords: Levonorgestrel-Releasing Intrauterine Device; Menstrual Cycle Phase; Ovarian Cyst
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early Follicular Phase: LNG-IUD inserted during early follicular phase (days 1-5).
- Late Follicular Phase: LNG-IUD inserted during late follicular phase (days 6-13).
- Early Luteal Phase: LNG-IUD inserted during early luteal phase (days 14-21).
- Late Luteal Phase: LNG-IUD inserted during late luteal phase (days 22-28).

SUMMARY:
In this prospective observational study, the effect of timing of insertion (early/late follicular; early/late luteal) on ovarian cyst development in women receiving an LNG-IUD will be assessed ultrasonographically at months 0, 3, 6, and 12. Secondary outcomes include cyst size/structure, bleeding pattern, pain, and other adverse events.

DETAILED DESCRIPTION:
The menstrual cycle will be divided into four subphases, and the LNG-IUD will be placed according to these phases.Participants will be assessed initially with a gynecological examination, ultrasound, and hormone profile (FSH, LH, TSH, prolactin, estradiol, progesterone); they will be followed up with ultrasound at months 0, 3, 6, and 12.There is no randomization or blinding (observational design).Data analysis will be conducted using chi-square/Fisher, with Yates correction if necessary, and Cramer's V/phi as the effect size (p<0.05/0.01).

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age: 18-45 years
* Patients with indications for LNG-IUD (levonorgestrel-containing intrauterine device) insertion (abnormal uterine bleeding, menorrhagia, dysmenorrhea, endometriosis, adenomyosis, hormonally induced dysfunctional uterine bleeding, endometrial protection in women receiving postmenopausal hormone replacement therapy, and endouterine hyperplasia without atypia)
* Patients without contraindications for LNG-IUD (no suspected pregnancy, no serious uterine anomalies (Müllerian anomalies), no active pelvic infection, no history of serious liver disease or breast cancer, and no anatomical or clinical contraindications to IUD insertion) will be included.
* They must not have used oral contraceptives for at least 3 months.
* The previous IUD must have been removed at least 1 year prior.
* Those who signed the informed consent form and agreed to participate voluntarily will be included in the study.
* Those who have not used steroidal anti-inflammatory drugs within 24 hours of insertion of a levonorgestrel-containing IUD will be included in the study.

Exclusion Criteria:

* Pregnancy history or current pregnancy
* Patients using hormone therapy
* Patients with adnexal masses
* Patients with severe systemic diseases (uncontrolled diabetes, advanced cardiovascular disease, active malignancies (especially hormone-sensitive ones), advanced liver or kidney failure, systemic connective tissue diseases)
* Patients with contraindications to the levonorgestrel IUD (suspected pregnancy, severe uterine anomaly, active pelvic infection, severe liver disease, or a history of breast cancer, anatomical or clinical obstacles to intrauterine device insertion)
* Patients with psychological disabilities
* Patients who refuse to sign the informed consent form
* Patients who cannot be followed up will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of women aged 18 to 45 years who are clinically indicated for levonorgestrel-releasing intrauterine device (LNG-IUD) insertion for contraception or therapeutic purposes. Participants will be recruited from the outpatient gynecology clinic of SBÜ Gaziosmanpaşa Training and Research Hospital.
  All participants will have regular menstrual cycles and no contraindications to LNG-IUD use. They will be assigned to one of four observational cohorts (early follicular, late follicular, early luteal, or late luteal phase) according to the menstrual phase at the time of insertion.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ovarian Cyst Formation | Baseline, 3 months, 6 months, and 12 months post-insertion
  Occurrence of new ovarian cysts detected by transvaginal or transabdominal ultrasound after LNG-IUD insertion.

CONTACTS AND LOCATIONS:
Overall Officials: havva betül bacak, md, Principal Investigator — SBÜ Gaziosmanpaşa Training and Research Hospital
Locations (1):
- SBÜ Gaziosmanpaşa Training and Research Hospital, Gaziosmanpaşa, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No